### **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT03693430 |
| Sponsor trial ID: | NN9536-4378 |
| Official title of study: | Two-year effect and safety of semaglutide 2.4 mg once-weekly in subjects with overweight or obesity |
| Document date*: | 12 April 2021 |

<sup>\*</sup>Document date refers to the date on which the document was most recently updated.

Note: The date in the header from Page 2 is the date of compilation of the documents and not of an update to content.

| Semaglutide s.c. 2.4 mg once weekly | | Date: | 11 May 2021 | Novo Nordisk |
|---|---|---|---|---|
| Trial ID: NN9536 4378 | CONFIDENTIAL | Version: | 1.0 | I |
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | I |
| Appendix 16.1.9 | | | | I |

### 16.1.9 Documentation of statistical methods

### List of contents

Statistical analysis plan Link

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 12 April 2021 | **Novo Nordisk**1.0
Final

Statistical Analysis Plan

**Trial ID: NN9536-4378** 

### STEP 5

Two-year effect and safety of semaglutide 2.4 mg onceweekly in subjects with overweight or obesity

Redacted statistical analysis plan Includes redaction of personal identifiable information only.

Author

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page:

1.0 Final


12 April 2021 | Novo Nordisk

### **Table of contents**

| | | | | | Page |
|---|---|---|---|---|---|
| Ta | ble of o | contents | | | 2 |
| Li | st of ab | breviation | ıs | | 3 |
| 1 | Intro | duction | | | 4 |
| | 1.1 | Trial in | formation | | 4 |
| | | 1.1.1 | Objective | (s) | 4 |
| | | | 1.1.1.1 | Primary objective | 4 |
| | | | 1.1.1.2 | Secondary objectives | 4 |
| | | 1.1.2 | Estimands | 3 | 4 |
| | | | 1.1.2.1 | Primary estimand | |
| | | | 1.1.2.2 | Secondary estimand | 4 |
| | | 1.1.3 | Endpoints | S | 5 |
| | | | 1.1.3.1 | Primary endpoint | 5 |
| | | | 1.1.3.2 | Secondary endpoints | 5 |
| | | 1.1.4 | Type of tr | ial | 6 |
| | 1.2 | Scope o | of the statistica | al analysis plan | 7 |
| 2 | Static | stical cons | iderations | | 7 |
| _ | 2.1 | | | nation | |
| | 2.2 | | | s sets | |
| | 2.3 | | • | 5005 | |
| | 2.5 | 2.3.1 | | ndpoint | |
| | | 2.3.2 | • | y endpoints | |
| | | 21312 | 2.3.2.1 | · | |
| | | | 2.3.2.2 | Supportive secondary endpoints | |
| | | 2.3.3 | | ry endpoints | |
| | | 2.0.0 | 2.3.3.1 | • | |
| | | 2.3.4 | | ve statistical analysis for pharmacogenetics and biomarkers | |
| | | 2.3.5 | | lyses | |
| | 2.4 | | | or pharmacodynamic modelling | |
| 3 | Chan | ges to the | statistical an | alyses planned in the protocol | 21 |
| | 3.1 | Trial-sp | ecific change | S | 21 |
| | 3.2 | Change | s applied acro | oss STEP trials | 22 |
| 4 | Chan | ge log | | | 24 |
| _ | D 6 | _ | | | 2.7 |

Statistical Analysis Plan

Date: 12 April 2021 Novo Nordisk

Trial ID: NN9536 4378

Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


 Version:
 1.0

 Status:
 Final

 Page:

### List of abbreviations

AD available but discontinued

AE adverse event

ANCOVA analysis of covariance

AT available on randomised treatment

BMI body mass index
CI confidence interval
dBP diastolic blood pressure

FAS full analysis set FFA free fatty acid

FPG fasting plasma glucose
HbA1c glycated haemoglobin
HDL high density lipoprotein

hsCRP high-sensitivity C-Reactive Protein

LAO-OT last available observation during the on-treatment period

LDL low-density lipoprotein

MD missing and discontinued

MedDRAMedical Dictionary for Regulatory ActivitiesMMRMmixed model for repeated measurements

MT missing on randomised treatment

OR odds ratio

PYE patient years of exposure
PYO patient years of observation

RD-MI multiple imputation using retrieved subjects

SAE serious adverse event
SAP statistical analysis plan
SAS safety analysis set
sBP systolic blood pressure

s.c. subcutaneus
SD standard deviation

TEAE treatment-emergent adverse event VLDL very low density lipoprotein

WC waist circumference

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 12 April 2021 1.0 Final


Novo Nordisk

### 1 Introduction

#### 1.1 Trial information

### 1.1.1 Objective(s)

### 1.1.1.1 Primary objective

To compare the two-year effect of semaglutide s.c. 2.4 mg once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with overweight or obesity on body weight.

### 1.1.1.2 Secondary objectives

To compare the two-year effect of semaglutide s.c. 2.4 mg once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with overweight or obesity on:

- Cardiovascular risk factors
- Glucose metabolism

To compare the one-year effect of semaglutide s.c. 2.4 mg once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with overweight or obesity on body weight.

To compare the two-year safety and tolerability of semaglutide s.c. 2.4 mg once weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with overweight or obesity.

#### 1.1.2 Estimands

#### 1.1.2.1 Primary estimand

The estimand will quantify the average treatment effect of semaglutide relative to semaglutide placebo after 104 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects regardless of adherence to treatment and regardless of initiation of other anti-obesity therapies (i.e. weight management drugs or bariatric surgery) ("treatment policy" estimand). The estimand will cover all effect-related objectives.

The following expansion of the primary estimand will cover the supportive secondary objectives related to body weight. The estimand will quantify the average treatment effect of semaglutide relative to semaglutide placebo after 52 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects regardless of adherence to treatment and regardless of initiation of other anti-obesity therapies.

### 1.1.2.2 Secondary estimand

The estimand will quantify the average treatment effect of semaglutide relative to semaglutide placebo after 104 weeks, as an adjunct to a reduced-calorie diet and increased physical activity, in all randomised subjects had they remained on their randomised treatment for the entire planned duration of the trial and not initiated any other anti-obesity therapies (i.e. weight management drugs

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page:

12 April 2021 | Novo Nordisk Final


or bariatric surgery) ("hypothetical" estimand). The estimand will cover all effect-related objectives.

#### 1.1.3 **Endpoints**

#### 1.1.3.1 Primary endpoint

The primary endpoints addressing the primary objective:

- Change from baseline (week 0) to week 104 in body weight (%)
- Subjects who after 104 weeks achieve (yes/no):
  - Body weight reduction  $\geq 5\%$  from baseline (week 0)

#### 1.1.3.2 **Secondary endpoints**

The confirmatory and supportive secondary endpoints addressing the primary and secondary objectives are listed below.

### Confirmatory secondary endpoints

- Subjects who after 104 weeks achieve (yes/no):
  - Body weight reduction  $\geq 10\%$  from baseline (week 0)
  - Body weight reduction  $\geq 15\%$  from baseline (week 0)
- Change from baseline (week 0) to week 104 in:
  - Waist circumference (cm)
  - Systolic blood pressure (mmHg)

### Supportive secondary endpoints

Effect endpoints:

- Change from baseline (week 0) to week 104 in:
  - Body weight reduction  $\geq 20\%$  from baseline (week 0)
  - Body weight (kg)
  - BMI  $(kg/m^2)$
  - HbA<sub>1c</sub> (%, mmol/mol)
  - FPG (mg/dL, mmol/L)
  - Fasting serum insulin (mIU/L, pmol/L)
  - Diastolic blood pressure (mmHg)
  - Lipids (mg/dL, mmol/L)
    - Total cholesterol
    - High density lipoprotein (HDL) cholesterol
    - Low density lipoprotein (LDL) cholesterol
    - Very low density lipoprotein (VLDL) cholesterol
    - Free fatty acids (FFA)
    - Triglycerides
    - High sensitivity C-Reactive Protein (hsCRP) (mg/L)
- Change from baseline (week 0) to week 52 in:
  - Body weight (%, kg)

 Statistical Analysis Plan
 Date:
 12 April 2021
 Novo Nordisk

 Trial ID: NN9536-4378
 Version:
 1.0
 1.0

 UTN:U1111-1202-1740
 Status:
 Final

 EudraCT No.:2017-003726-32
 Page:

- BMI  $(kg/m^2)$
- Waist circumference (cm)
- Subjects who after 52 weeks achieve (yes/no):
  - Body weight reduction  $\geq 5\%$  from baseline (week 0)
  - Body weight reduction  $\geq 10\%$  from baseline (week 0)
  - Body weight reduction  $\geq 15\%$  from baseline (week 0)
  - Body weight reduction  $\geq 20\%$  from baseline (week 0)

### Safety endpoints:

- Number of treatment emergent adverse events (TEAEs) from baseline (week 0) to week 111
- Number of serious adverse events (SAEs) from baseline (week 0) to week 111
- Change from baseline (week 0) to week 104 in:
  - Pulse (bpm)
  - Amylase (U/L)
  - Lipase (U/L)
  - Calcitonin (ng/L)

### **Exploratory endpoints**

The exploratory endpoints addressing the exploratory objectives:

- Change from baseline (week 0) to week 104 in:
  - Glycaemic category (normo-glycaemia, pre-diabetes, T2D)
  - Antihypertensive medication (decrease, no change, increase)
  - Lipid-lowering medication (decrease, no change, increase)
- Subjects who from randomisation to week 104 have permanently discontinued randomised trial product (yes/no)
- Time to permanent discontinuation of randomised trial product (weeks)
- Control of Eating Questionnaire (CoEQ): Scores from the 4 domains and 19 individual items (applicable for US and Canada only)

### 1.1.4 Type of trial

This is a 104-week, randomised, double-blind, placebo-controlled, two-armed, parallel group, multi-centre, multinational clinical trial comparing semaglutide 2.4 mg once weekly with semaglutide placebo, as an adjunct to a reduced-calorie diet and increased physical activity, in subjects with overweight or obesity.

The trial includes a screening visit to assess the subject's eligibility followed by visits/phone contacts every 2<sup>nd</sup> week during dose escalation. From week 20, visits/phone contacts will take place every 4<sup>th</sup> week for the remaining maintenance period until end of treatment (week 104). A follow-up visit ('End of trial') for safety assessments is scheduled 7 weeks after end of treatment to account for the exposure to the long half-life of semaglutide.

### 1.2 Scope of the statistical analysis plan

This statistical analysis plan (SAP) is based on the protocol for trial NN9536-4378 "Two-year effect and safety of semaglutide 2.4 mg once-weekly in subjects with overweight and obesity", version 3.0 (29 June 2018) as well as amendment 1, and includes more detailed procedures for executing the statistical analyses of the primary and secondary endpoints. Statistical analyses and a number of clarifications additional to those specified in the trial protocol are pre-specified with this SAP. All changes to the statistical analyses planned in the trial protocol are documented in section 3.

### 2 Statistical considerations

#### Taxonomy of week 104 assessments

For each subject a given assessment at week 104 may be available or missing and Table 2-1 describes the taxonomy for this. Note, this is done per assessment and per subject; subjects may be a different type for different assessments (a subject may have "available on randomised treatment (AT)" for body weight but "missing on randomised treatment (MT)" for waist circumference).

Table 2-1 Taxonomy for subjects based on week 104 assessments

| Assessment<br>at week 104 | Subjects on<br>randomised<br>treatment at<br>week 104 | Type description | Type<br>Abbreviation |
|---|---|---|---|
| Available | Yes | Available on randomised treatment: Subjects who complete the trial on randomised treatment with an assessment at week 104: Includes those that stop and restart trial product. | AT |
| | No | Available but discontinued Subjects who discontinued randomised treatment prematurely but returned to have an assessment at week 104. These are also called retrieved subjects | AD |
| Missing | Yes | Missing on randomised treatment: Subjects who complete the trial on randomised treatment without an assessment at week 104: Includes those that stop and restart trial product. | MT |
| | No | Missing and discontinued: Subjects who discontinued randomised treatment prematurely and did not return to have an assessment at week 104. These are also called non-retrieved subjects | MD |

#### 2.1 Sample size determination

The sample size was primarily defined to ensure sufficient power for the two primary endpoints. Given the trial sample size, the power of statistical tests for all confirmatory endpoints is described below.

The tests of superiority of semaglutide 2.4 mg to semaglutide placebo for the primary and confirmatory secondary endpoints are performed using the fixed-sequence statistical strategy. This strategy tests the endpoints using a predefined hierarchical order, all at the significance level of 5%, moving to test the next endpoint only after a statistically significant superiority result (p-value < 5%) on the previous endpoint. The test hierarchy is given in Table 2-2 with underlying assumptions, marginal power and effective power. The effective power is calculated under the assumption of independence of endpoints by multiplying the respective marginal powers successively. As the two primary endpoints are included in the statistical testing hierarchy,

| Statistical Analysis Plan<br>Trial ID: NN9536-4378<br>UTN:U1111-1202-1740<br>EudraCT No.:2017-003726-32 | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 12 April 2021<br>1.0<br>Final<br>8 of 25 | Novo Nordisk |
|---|---|---|---|---|
|---|---|---|---|---|

significant superiority of semaglutide 2.4 mg vs. semaglutide placebo must be demonstrated for each of the primary endpoints.

In the analysis approach addressing the primary estimand, week 104 assessments from retrieved subjects (AD) are used. These data are also used to impute missing measurements at week 104 for non-retrieved subjects (MD). The imputation is done separately within each treatment arm (see description below). However, for the power calculations missing values (MT and MD), regardless of treatment arm, are assumed to be similar to semaglutide placebo subjects. These assumptions are likely conservative with respect to the power, and correspond to the jump to reference sensitivity analysis planned below.

### **Assumptions**

The common assumptions for the power calculations are

- The significance level is 5%
- The randomisation ratio is 1:1
- For continuous endpoints the t-test on the mean difference assuming equal variances is used
- For binary endpoints the Pearson chi-square test for two independent proportions is used
- 40% of subjects discontinue permanently and 50% of these are retrieved (AD) at week 104
- All subjects in the semaglutide placebo arm are assumed to have same effect as subjects who complete the trial on semaglutide placebo (AT)
- Retrieved subjects (AD) in the semaglutide 2.4 mg arm are assumed to have an effect corresponding to 25% of the treatment difference (compared to semaglutide placebo) of subjects who complete the trial on semaglutide 2.4 mg (AT)
- Non-retrieved subjects (MD) in the semaglutide 2.4 mg arm are assumed to have an effect corresponding to semaglutide placebo

Further assumptions made to calculate the power for each of the primary and confirmatory secondary endpoints are based on findings from other projects conducted by Novo Nordisk (NN8022 (SCALE), NN9535 (SUSTAIN), NN9924 (PIONEER)), and trial NN9536-4153 and are presented in Table 2-2. For weight, waist circumference and systolic blood pressure a 2 year completer was assumed to have 90% the effect of a 1 year completer.

Given these assumptions, the sample size of 300 subjects (150 in each arm), gives an effective power (marginal powers multiplied) of 43%. As sample size is primarily driven by the two primary endpoints, additional scenarios for assumptions are not included due to the high power for these endpoints.

| Statistical Analysis Plan | 1 | Date: | 12 April 2021 | Novo Nordisk |
|---|---|---|---|---|
| Trial ID: NN9536-4378 | CONFIDENTIAL | Version: | 1.0 | |
| UTN:U1111-1202-1740 | CONFIDENTIAL | Status: | Final | |
| EudraCT No.:2017-003726-32 | | Page: | 9 of 25 | |

Table 2-2 Assumptions, marginal power and effective power for each endpoint in the hierarchical testing procedure given an anticipated number of 300 randomised subjects

| Order | Endpoint | | ean (±SD) or<br>or completers<br>Semaglutide<br>placebo | Expected mean (±SD) or proportion Semaglutide 2.4 mg | Expected difference or proportion ratio | Marginal power (%) | Effective power (%) |
|---|---|---|---|---|---|---|---|
| 1 | % weight change # | 12.6 (±11) | 3.0 (±11) | 9.2 (±12) | 6.2%-points | > 99 | > 99 |
| 2 | 5% responders | 76% | 43% | 64% | 1.5 | 96 | 96 |
| 3 | 10% responders | 59% | 26% | 48% | 1.8 | 97 | 93 |
| 4 | 15% responders | 41% | 14% | 31% | 2.2 | 96 | 89 |
| 5 | WC change (cm) # | 9.3 (±11) | 4 (±11) | 7.4 (±12) | 3.4 cm | 69 | 62 |
| 6 | sBP change (mmHg) # | 7.6 (±13) | 1.5 (±13) | 5.5 (±14) | 4 mmHg | 69 | 43 |

SD = standard deviation; WC = waist circumference; sBP = systolic blood pressure; # shown as a positive number All tests in the hierarchy are based on the primary estimand

### 2.2 Definition of analysis sets

Two analysis sets are defined:

- The *full analysis set* (FAS) includes all randomised subjects according to the intention-to-treat principle. Subjects in the FAS will contribute to evaluation "as randomised".
- The *safety analysis set* (SAS) includes all randomised subjects exposed to at least one dose of randomised treatment. Subjects in the SAS will contribute to evaluation "as treated".

Any observation excluded from the analysis will be documented before database lock with the reason for exclusion provided.

Two observation periods are defined for each subject:

- In-trial: The *in-trial period* is defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.
- On-treatment (with trial product): A time-point is considered as 'on-treatment' if any dose of trial product has been administered within the prior 2 weeks (14 days). The *on-treatment period* is defined as all times which are considered on-treatment.
  - In general, the on-treatment period will therefore be from the date of first trial product administration to date of last trial product administration (±14 days) excluding potential off-treatment time intervals triggered by at least two consecutive missed doses.
  - For the evaluation of adverse events, the lag time for each on-treatment time interval is 7 weeks (49 days).

The in-trial and on-treatment periods define the patient years of observation (PYO) and patient years of exposure (PYE), respectively, as the total time duration in the periods.

### 2.3 Statistical analyses

If necessary, a statistical analysis plan (SAP) may be written in addition to the protocol, including a more technical and detailed elaboration of the statistical analyses. The SAP will be finalised before database lock.

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status:

12 April 2021 | Novo Nordisk Final

Effect endpoints will be analysed using the FAS; safety endpoints will be analysed using the SAS.

Results from statistical analyses will generally be accompanied by two-sided 95% confidence intervals and corresponding p-values. Superiority will be claimed if p-values are less than 5% and the estimated treatment contrasts favours semaglutide 2.4 mg.

### Handling of missing baseline data

The last available and eligible observation at or before randomisation, is used as the baseline value. If no assessments are available, the mean value at randomisation across all subjects is used as the baseline value.

#### 2.3.1 **Primary endpoint**

Definition of primary endpoint: % weight change

Change from baseline (week 0) to week 104 in body weight (%) is defined as

% weight change = 
$$\frac{\text{(body weight at week } 104 - body weight at baseline)}}{\text{body weight at baseline}} \times 100.$$

Definition of primary endpoint: 5% responders

A body weight reduction of at least 5% from baseline (week 0) to week 104 is defined as

5% responder = 
$$\begin{cases} 1 & \text{if } \% \text{ weight change} \le -5\% \\ 0 & \text{if } \% \text{ weight change} > -5\% \end{cases}$$

#### Analyses addressing the primary estimand

The following statistical analyses and imputation methods are designed to address the primary estimand, i.e. to assess the effectiveness of semaglutide 2.4 mg.

The analysis model for % weight change is a linear regression (ANCOVA) of % weight change with randomised treatment as a factor and baseline body weight (kg) as covariate. The estimated treatment difference between semaglutide 2.4 mg and semaglutide placebo will be reported together with the associated two-sided 95% CI and corresponding p-value.

The analysis model for the 5% responder endpoint is a logistic regression using randomised treatment as a factor and baseline body weight (kg) as covariate. The estimated odds ratio (OR) between semaglutide 2.4 mg and semaglutide placebo will be reported together with the associated two-sided 95% CI and corresponding p-value.

The superiority tests of semaglutide 2.4 mg vs. semaglutide placebo will be carried out as follows for the two analysis models.

Let μ<sub>semaglutide</sub> and μ<sub>semaglutide placebo</sub> denote the true mean of % weight change for semaglutide 2.4 mg and semaglutide placebo group, respectively. The null and alternative hypotheses tested are

H: 
$$\mu_{semaglutide} \ge \mu_{semaglutide \ placebo} \ vs$$
  
 $H_A$ :  $\mu_{semaglutide} < \mu_{semaglutide \ placebo}$ .

The hypothesis will be rejected and superiority claimed, if the upper limit of the estimated two-sided 95% CI is below 0.

Let OR<sub>semaglutide/semaglutide placebo</sub> denote the true odds ratio between semaglutide 2.4 mg and semaglutide placebo. The null and alternative hypotheses tested are

 $H: OR_{semaglutide/semaglutide\ placebo} \le 1\ vs$  $H_A: OR_{semaglutide/semaglutide\ placebo} > 1.$ 

The hypothesis will be rejected and superiority claimed, if the lower limit of the estimated two-sided 95% CI is above 1.

Handling of missing week 104 values for the primary estimand

All available data at week 104 (AT and AD) are used and missing values (MT and MD) at week 104 will be imputed and the endpoints will be derived from the imputed values. Several approaches for imputation will be applied. First, a description of the primary imputation approach to address the primary estimand for the primary endpoints is given followed by a description of the sensitivity analyses used to assess the robustness of the primary analysis results. The sensitivity analyses investigate how assumptions on body weight development after discontinuation of randomised treatment impact the estimated treatment contrasts between semaglutide 2.4 mg and semaglutide placebo. An illustration of all imputation approaches for the primary estimand is given in Figure 1.

### Primary imputation approach for the primary estimand

Multiple imputation approach using retrieved subjects (RD-MI): The primary imputation approach for the primary estimand is a multiple imputation similar to the one described by McEvoy1. Missing body weight measurement at week 104 for non-retrieved subjects (MD) are imputed using assessments from retrieved subjects (AD) in each randomised treatment arm. This will be done according to the timing of last available observation on-treatment (LAO-OT) of body weight prior to week 104. Missing body weight measurements at week 104 for subjects on randomised treatment (MT) are imputed in a similar way by sampling from available measurements at week 104 from subjects on randomised treatment (AT) in the relevant randomised treatment arm. The multiple imputation approach is done in three steps:

1. **Imputation**: Defines an imputation model using retrieved subjects (AD) from FAS and done within groups defined by randomised treatment and the timing of the LAO-OT of body weight. The model will be a linear regression of body weight (kg) at week 104 with gender (male/female), baseline BMI (kg/m²) (in categories -<35, 35-<40, ≥40) and timing of the LAO-OT of body weight as factors and baseline body weight (kg) and LAO-OT of body weight (kg) as covariates. No interactions will be included. The grouping of timing will be done by quarters (intervals of 26 weeks for endpoints evaluating the change after 104 weeks, intervals of 13 weeks for endpoints evaluating the change after 52 weeks). If timing by quarters is too restrictive, halves (intervals of 52 weeks for endpoints evaluating the change after 52 weeks) or excluding timing will be used. The timing by quarters or halves is defined as too restrictive if the imputation model cannot be fit due to inadequate numbers of retrieved subjects in 1 or more groups. If the imputation model still cannot be fit after excluding timing then the model will be further reduced

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: 2 April 2021 1.0 Final 12 of 25

12 April 2021 | Novo Nordisk

until the model can be fit. Reduction will be done in a fixed order by first removing gender, then collapsing the two highest baseline BMI groups into one (≥35) and finally removing baseline BMI group. If no LAO-OT exists post-baseline then LAO-OT will be the baseline body weight and the timing will be the first interval. If any subjects are MT, an imputation model for missing body weight measurements at week 104 for MT subjects will also be defined using AT subjects in a similar way. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 104 body weight values for each randomised treatment arm. This will be done 1,000 times and results in 1,000 complete data sets.

- 2. **Analysis**: Analysis of each of the 1,000 complete data sets, using the analysis models (ANCOVA and logistic regression) results in 1,000 times 2 estimations.
- 3. **Pooling**: Integrates the 1,000 times 2 estimation results into two final results using Rubin's formula.

Based on NN9536-4153 phase 2 results 1,000 copies should be sufficient to establish stable results. If 1,000 copies are insufficient, 10,000 copies will be used. The multiple imputations will be generated using Novo Nordisk trial number 95364378 as seed number. In addition to the seed number, it is specified that the dataset is sorted by subject ID.

### Sensitivity analyses

Jump to reference multiple imputation approach (J2R-MI): Missing values of body weight at week 104 (MT and MD) for both the semaglutide 2.4 mg and semaglutide placebo group are imputed by sampling among all available assessments at week 104 in the semaglutide placebo group (AT and AD). This approach makes the assumption that subjects instantly after discontinuation lose any effect of randomised treatment beyond what can be expected from semaglutide placebo treatment as adjunct to reduced-calorie diet and increased physical activity2. The multiple imputation approach is done as above with the first step replaced by:

1. **Imputation**: Defines an imputation model using semaglutide placebo subjects from FAS with a week 104 measurement (AT and AD). The model will be a linear regression of body weight (kg) at week 104 with gender (male/female), BMI (kg/m²) (in categories -<35, 35-<40, ≥40) as factors and baseline body weight (kg) as covariate. No interactions will be included. If the imputation model cannot be fit due to inadequate numbers of retrieved subjects in one or more groups, then the imputation model will be reduced until the model can be fit. Reduction will be done in a fixed order by first removing gender, then collapsing the two highest baseline BMI groups into one (≥35) and finally removing baseline BMI group. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 104 body weight values for each randomised treatment arm. This will be done 1,000 times and results in 1,000 complete data sets.

The jump to reference approach is the basis for the sample size calculations.

A single imputation approach as done by Sacks3 (S1-SI and S2-SI): Missing weight measurements at week 104 for non-retrieved subjects (MD) are imputed using a weight regain rate of 0.3 kg/month after LAO but truncated at no change from baseline whenever the extrapolation would lead to a positive weight gain relative to baseline. If a subject's weight at drug discontinuation represented a

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 12 April 2021 1.0 Final 13 of 25

Novo Nordisk

gain in weight relative to baseline, no additional gain will be imputed, and the unfavourable gain is carried forward to week 104. The weight regain imputation will be done for both randomised arms (S1-SI). Additionally, a version where only the semaglutide 2.4 mg arm uses the regain rate while the semaglutide placebo arm uses last available observation (corresponding to a weight regain rate of 0 kg/month) will be performed (S2-SI). For both versions, missing weight measurements at week 104 for subjects on randomised treatment (MT) are imputed by using LAO.

Tipping-point multiple imputation analysis (TP-MI): First, missing data are imputed according to the primary multiple imputation approach. Then, a penalty is added to the imputed values at week 104. The approach is to explore a range of penalties for both treatment groups, and the impact these would have on the study conclusions. The 2-dimensional space of penalties covering the range from -30% to 30% will be explored for both treatment groups. This sensitivity analysis evaluates the robustness of the superiority conclusions to departures from the observed change in body weight in both treatment groups.

Mixed model for repeated measurements (MMRM): This 'MMRM for effectiveness' will use all assessments regardless of adherence to randomised treatment, including assessments at week 104 for retrieved drop-outs (AD). The MMRM for effectiveness will be fitted using the same factor and covariate as for the primary analyses all nested within visit. An unstructured covariance matrix for measurements within the same subject will be employed, assuming that measurements for different subjects are independent. For the 5% responder analysis, the same MMRM will be applied except that body weight (kg) will be used as response variable in the model. Individual missing values for body weight at week 104 will be predicted from the MMRM and used to classify each subject as 5% responder or not. This classification will then be analysed using the same logistic regression model as in the primary analysis of the primary estimand.

Subjects with missing week 104 assessment as non-responders: For the 5% responder analysis an analysis using subjects with missing week 104 assessment as non-responders in the logistic regressions will be done.

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page:

12 April 2021 1.0 Final 14 of 25

Novo Nordisk



Figure 1 Illustration of imputation approaches for the primary estimand

### Analysis addressing the secondary estimand

The secondary estimand for % weight change addresses the efficacy of semaglutide 2.4 mg and will be assessed using a 'MMRM for efficacy'. Week 104 assessments for retrieved drop-outs (AD) are not used in this analysis. The MMRM for efficacy will use assessments only from subjects who are taking the randomised treatment until end of treatment or until first discontinuing of randomised treatment. The derived date of the second consecutive missed dose will be used as the latest date for using assessments in this MMRM. The assessment closest in time and before the derived date of the

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: 2 April 2021 1.0 Final 15 of 25

12 April 2021 | Novo Nordisk

second consecutive missed dose will be used as last assessment on randomised treatment. For subjects who initiate other anti-obesity therapies before completion or first discontinuing of randomised treatment, the date of starting weight management drugs or undergoing bariatric surgery will be used as latest date for using assessments in this MMRM. Similarly, the assessment closest in time and before the date of starting weight management drugs or undergoing bariatric surgery will be used as last assessment on randomised treatment. The MMRM for efficacy will be fitted using % weight change and the same factor and covariate as for the primary analyses all nested within visit. An unstructured covariance matrix for measurements within the same subject will be employed, assuming that measurements for different subjects are independent.

The secondary estimand for 5% responders will be assessed using the same MMRM for efficacy except that body weight (kg) will be used as response variable in the model. For subjects with missing body weight at week 104, individual values for body weight will be predicted from the MMRM and used to classify each subject as 5% responder or not. This classification will then be analysed using a logistic regression model with treatment as the only factor.

An overview of all analysis and imputation methods to address the primary and secondary estimands for the primary endpoints is given in Table 2-3.

### 2.3.2 Secondary endpoints

### 2.3.2.1 Confirmatory secondary endpoints

Confirmatory secondary endpoints are listed in section 4.2.2.1 of the study protocol and are all included in the fixed-sequence statistical strategy, see above. All tests are tests of superiority of semaglutide 2.4 mg to semaglutide placebo.

### Analyses addressing the primary estimand

All confirmatory secondary endpoints will be analysed using the same imputation approach as used for the primary endpoints and to address the primary estimand. The imputation model is the same as for the primary endpoints with body weight replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % weight change with baseline body weight replaced by the baseline assessment of the endpoint to be analysed. The statistical model for body weight responder endpoints will be logistic regression with factors and covariate as for the primary endpoint 5% responders.

#### Analyses addressing the secondary estimand

The confirmatory secondary endpoints which relate to the primary objective for week 104 will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoints.

Sensitivity analyses for confirmatory secondary endpoints

For all continuous confirmatory secondary endpoints a sensitivity analysis using jump to reference as imputation approach will be carried out. For all binary confirmatory secondary endpoints a sensitivity analysis using non-retrieved subjects as non-responders will be carried out.

| Statistical Analysis Plan Date: 12 April 2021 Novo N | 0: NN9536-4378<br>1111-1202-1740 |
|---|---|
|---|---|

An overview of all analysis and imputation methods to address the primary and secondary estimands for confirmatory secondary endpoints is given in Table 2-3.

Table 2-3 Analysis and imputation methods to address the primary and secondary estimands for the primary and confirmatory secondary endpoints in the statistical testing hierarchy

| Objective | Endpoint | Test<br>order | Endpoint<br>type | Estimand | Analysis<br>set | Statistical<br>model | Imputation approach | Sensitivity analyses |
|---|---|---|---|---|---|---|---|---|
| Primary en | dpoints | • | | | | - | | |
| Primary | % weight change | 1 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI<br>S1-SI<br>S2-SI<br>TP-MI<br>MMRM |
| | | | | Secondary | FAS | MMRM | - | - |
| Primary | 5% responders | 2 | Binary | Primary | FAS | LR | RD-MI | J2R-MI<br>S1-SI<br>S2-SI<br>TP-MI<br>MMRM<br>Non-<br>responder |
| | | | | Secondary | FAS | LR | MMRM | - |
| Confirmato | ry secondary endpoints | | | | | | | |
| Primary | 10% responders | 3 | Binary | Primary | FAS | LR | RD-MI | Non-<br>responders |
| | | | | Secondary | FAS | LR | MMRM | - |
| Primary | 15% responders | 4 | Binary | Primary | FAS | LR | RD-MI | Non-<br>responders |
| | | | | Secondary | FAS | LR | MMRM | - |
| Primary | WC change (cm) | 5 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI |
| | | | | Secondary | FAS | MMRM | - | - |
| Secondary | sBP change (mmHg) | 6 | Continuous | Primary | FAS | ANCOVA | RD-MI | J2R-MI |
| | | | | Secondary | FAS | MMRM | - | |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; J2R-MI = jump to reference multiple imputation; S1-SI and S2-SI = single imputation as done by Sacks; TP-MI = tipping point multiple imputation; MMRM = mixed model for repeated measurements; LR = logistic regression; WC = waist circumference; sBP = systolic blood pressure

Test order refers to the order of the endpoint in the statistical test hierarchy outlined in Table 2-3.

### 2.3.2.2 Supportive secondary endpoints

Supportive secondary endpoints are listed in section 4.2.2.2 of the study protocol. All tests are tests of superiority of semaglutide 2.4 mg to semaglutide placebo.

### Analyses addressing the primary estimand

The effect-related supportive secondary endpoints will be analysed using the same imputation approach as used for the primary endpoints and to address the primary estimand. The imputation model is the same as for the primary endpoints with body weight replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % weight change with baseline body weight replaced by the baseline assessment of the endpoint to be analysed.

For lipids, fasting serum insulin and hsCRP a multiplicative model will be used, i.e. the ratio between post randomisation measurements and baseline will be calculated instead of differences, and both the dependent variable and covariate will be log-transformed.

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 12 April 2021 1.0 Final 17 of 25

Novo Nordisk

### Analyses addressing the secondary estimand

The supportive secondary endpoints which relate to the primary objective will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoints.

### Additional considerations for statistical analyses

Supportive secondary endpoints evaluating the one-year effect of semaglutide 2.4 mg will be analysed using the same imputation approach as used for the primary endpoints and to address the primary estimand. The imputation model is the same as for the primary endpoints. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % weight change. The statistical model for body weight responder endpoints will be logistic regression with factor and covariate as for the primary endpoint 5% responders.

The supportive secondary endpoint "Change from baseline to week 52 in body weight (%)" will be compared to the primary endpoint "Change from baseline to week 104 in body weight (%)".

Sensitivity analyses for supportive secondary endpoints

For supportive secondary endpoints no sensitivity analysis will be carried out.

### Analysis of safety endpoints

The safety endpoint pulse will be analysed using an MMRM for efficacy as described in section 2.3.1. For amylase, lipase and calcitonin descriptive statistics will be provided. The analysis of calcitonin will be stratified by gender. Amylase, lipase and calcitonin will be log-transformed.

Adverse events will be defined as "treatment-emergent" (TEAE), if the onset of the event occurs in the on-treatment period (see definition in section 2.2). TEAEs and SAEs will be summarised by descriptive statistics, such as frequencies and rates. No formal statistical inference will be carried out based on the number of TEAEs and SAEs. All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA).

An overview of all analysis and imputation methods to address the primary and secondary estimands for supportive secondary endpoints is given in Table 2-4.

Table 2-4 Analysis and imputation methods to address the primary and secondary estimands for supportive secondary endpoints

| Objective | Endpoint | Endpoint | Estimand | Analysis | Statistical | Imputation | Sensitivity |
|---|---|---|---|---|---|---|---|
| - | | type | | set | model | approach | analyses |
| Supportive | secondary endpoints (effect related) | | | | | | |
| From baselin | ne to week 104 | | | | | | |
| Primary | 20% responders | Binary | Primary | FAS | LR | RD-MI | - |
| - | | | Secondary | FAS | LR | MMRM | - |
| Primary | Weight change (kg) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| - | | | Secondary | FAS | MMRM | - | - |
| Primary | BMI change (kg/m <sup>2</sup> ) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| - | | | Secondary | FAS | MMRM | - | - |
| Secondary | HbA <sub>1c</sub> change (%, mmol/mol) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| • | | | Secondary | FAS | MMRM | - | - |
| Secondary | FPG change (mg/dL, mmol/L) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| • | | | Secondary | FAS | MMRM | - | - |
| Secondary | Fasting serum insulin change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| • | (mIU/L, pmol/L) | | Secondary | FAS | MMRM | - | - |

Statistical Analysis Plan
Trial ID: NN9536-4378
UTN:U1111-1202-1740

Date: 12 April 2021 | Novo Nordisk
Version: 1.0
Status: Final

Page:


| Secondary | dBP change (mmHg) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
|---|---|---|---|---|---|---|---|
| - | | | Secondary | FAS | MMRM | - | - |
| Secondary | Total cholesterol change (mg/dL, | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| - | mmol/L) | | Secondary | FAS | MMRM | - | - |
| Secondary | HDL change (mg/dL, mmol/L) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| - | | | Secondary | FAS | MMRM | - | - |
| Secondary | LDL change (mg/dL, mmol/L) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Secondary | VLDL change (mg/dL, mmol/L) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Secondary | FFA change (mg/dL, mmol/L) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Secondary | Triglycerides change (mg/dL, | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | mmol/L) | | Secondary | FAS | MMRM | - | - |
| Secondary | hsCRP change (mg/L) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| - | | | Secondary | FAS | MMRM | - | - |
| From baselin | ne to week 52 | | | | | | |
| Secondary | Weight change (%, kg) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| - | | | Secondary | FAS | MMRM | - | - |
| Secondary | BMI change (kg/m²) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Secondary | WC change (cm) | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Secondary | 5% responders | Binary | Primary | FAS | LR | RD-MI | - |
| - | _ | | Secondary | FAS | LR | MMRM | - |
| Secondary | 10% responders | Binary | Primary | FAS | LR | RD-MI | - |
| | | | Secondary | FAS | LR | MMRM | - |
| Secondary | 15% responders | Binary | Primary | FAS | LR | RD-MI | - |
| | | | Secondary | FAS | LR | MMRM | - |
| Secondary | 20% responders | Binary | Primary | FAS | LR | RD-MI | - |
| - | | | Secondary | FAS | LR | MMRM | - |
| Supportive | secondary endpoints (safety related) | | | | | | |
| Secondary | Number of TEAEs | Continuous | - | SAS | - | - | - |
| Secondary | Number of SAEs | Continuous | - | SAS | - | - | - |
| Secondary | Pulse change (bpm) | Continuous | - | SAS | MMRM | - | - |
| Secondary | Amylase change (U/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Lipase change (U/L) | Continuous | - | SAS | Descriptive statistics | - | - |
| Secondary | Calcitonin change (ng/L) | Continuous | - | SAS | Descriptive statistics | - | - |

FAS = full analysis set; ANCOVA = analysis of covariance; RD-MI = multiple imputation using retrieved subjects; MMRM = mixed model for repeated measurements; BMI = body mass index; HbA<sub>1c</sub> = Hemoglobin A1c; FPG = fasting plasma glucose; dBP = diastolic blood pressure; HDL = high density lipoprotein; LDL = low density lipoprotein; VLDL = very low density lipoprotein; FFA = free fatty acids; hsCRP = high sensitivity C-Reactive Protein; WC = waist circumference; LR = logistic regression; TEAEs = treatment emergent adverse events; SAEs = serious adverse events

### 2.3.3 Exploratory endpoints

EudraCT No.:2017-003726-32

Exploratory endpoints are listed in 4.2.3 of the study protocol. Observed data for exploratory endpoints will be summarised by the descriptive statistics.

### 2.3.3.1 Control of Eating Questionnaire (CoEQ)

The CoEQ comprises 21-items designed to assess the intensity and type of food craving, as well as subjective sensations of appetite and mood4. In STEP5 a version with 19 items has been used (see Table 2-5). One of the two excluded items is open-ended and addresses specific foods, and the other excluded item concerns how difficult it has been to resist this specific food; and the items are therefore not part of any of the four domains.

Statistical Analysis Plan
Trial ID: NN9536-4378
UTN:U1111-1202-1740

Date: 12 April 2021 | Novo Nordisk
Version: 1.0
Status: Final

Page:


### Table 2-5 Overview of items in CoEQ

EudraCT No.:2017-003726-32

| Item<br>No. | Item text | Response scale |
|---|---|---|
| 1 | How hungry have you felt? | 10 = Extremely hungry, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all hungry |
| 2 | How full have you felt? | 10 = Extremely full, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all full |
| 3 | How strong was your desire to eat sweet foods? | 10 = Extremely strong, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all strong |
| 4 | How strong was your desire to eat salty and spicy foods (french fries, potato chips, burgers, pizza, etc.)? | 10 = Extremely strong, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all strong |
| 5 | How happy have you felt? | 10 = Extremely happy, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all happy |
| 6 | How anxious have you felt? | 10 = Extremely anxious, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all anxious |
| 6<br>7<br>8<br>9 | How alert have you felt? | 10 = Extremely alert, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all alert |
| 8 | How contented have you felt? | 10 = Extremely contended, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all contended |
| 9 | During the last 7 days how often have you had food cravings? | 10 = Very often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 10 | How strong have any food cravings been? | 10 = Extremely strong, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all strong |
| 11 | How difficult has it been to resist any food cravings? | 10 = Extremely difficult, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all difficult |
| 12 | How often have you eaten in response to food cravings? | 10 = After every one, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 13 | How often have you had cravings for chocolate and chocolate flavoured foods? | 10 = Extremely often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 14 | How often have you had cravings for other sweet foods (cakes, pastries, biscuits, etc)? | 10 = Extremely often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 15 | How often have you had cravings for fruit or fruit juice? | 10 = Extremely often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 16 | How often have you had cravings for dairy foods (cheese, yoghurt, milk, etc.)? | 10 = Extremely often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 17 | How often have you had cravings for starchy foods (bread, rice, pasta, etc.)? | 10 = Extremely often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 18 | How often have you had cravings for salty and spicy foods (french fries, potato chips, burgers, pizza, etc.)? | 10 = Extremely often, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all |
| 19 | Generally, how difficult has it been to control your eating? | 10 = Extremely difficult, 9, 8, 7, 6, 5, 4, 3, 2, 1, 0 = Not at all difficult |

### **Item scores**

The CoEQ item are scores on an 11-point graded response scale ranging from 10 to 0. No reversal of item scores will be done.

### **Domain scores**

The sum of the items in each domain is calculated, and divided by the number of items in the domain in order to obtain a domain score. Items 1 and 2 are not included in any domain score. Details are given in Table 2-6.

Table 2-6 Overview of domains for CoEQ

| Domain | Items included in domain | Comment |
|---|---|---|
| Craving Control | Question 9, 10, 11, 12 and 19 | The domain score is reversed such that a greater score |
| | | represents a greater level of Craving Control (i.e. 10 to 0, 9 to |
| | | 1,, 0 to 10) |
| Positive Mood | Question 5, 6, 7 and 8 | Scores from item 6 are reversed (i.e. 10 to 0, 9 to 1,, 0 to 10) |

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 12 April 2021 1.0 Final 20 of 25

Novo Nordisk

| Craving for Savoury | Question 4, 16, 17 and 18 |
|---------------------|----------------------------|
| Craving for Sweet | Question 3, 13, 14, and 15 |

Missing data at instrument level will be handled in the following way. To score a domain it is required that a least 50% of the items need to be answered. Then, the domain is scored based on the average of the items answered. If less than 50% of the items of a domain are answered no score will be derived.

Table 2-7 Analysis and imputation methods to address the primary and secondary estimands for exploratory endpoints

| Objective | Endpoint | Endpoint type | Estimand | Analysis set | Statistical model | Imputation approach | Sensitivity analyses |
|---|---|---|---|---|---|---|---|
| Exploratory endpo | nints | | ı | 1 | | | |
| From baseline to w | | | | | | | |
| Exploratory | CoEQ q1 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | I _ |
| Exploratory | COLQ q1 score change | Continuous | Secondary | FAS | MMRM | - | _ |
| Exploratory | CoEQ q2 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| | COLQ 42 score change | Commuous | Secondary | FAS | MMRM | - | _ |
| Exploratory | CoEQ q3 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| | COLQ do score change | | Secondary | FAS | MMRM | - | _ |
| Exploratory | CoEQ q4 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| 2p.ioravor) | Sez Q q. seere enunge | | Secondary | FAS | MMRM | - | _ |
| Exploratory | CoEQ q5 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | _ |
| <sub>7</sub> , | Q 4P 3 | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q6 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| 1 2 | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q7 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| 1 2 | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q8 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| 1 2 | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q9 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q10 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q11 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q12 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q13 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q14 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q15 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q16 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q17 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q18 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | CoEQ q19 score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | Craving Control score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |
| Exploratory | Positive Mood score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | |
| Exploratory | Craving for Savoury score | Continuous | Primary | FAS | ANCOVA | RD-MI | |
| | change | | Secondary | FAS | MMRM | - | - |
| Exploratory | Craving for Sweet score change | Continuous | Primary | FAS | ANCOVA | RD-MI | - |
| | | | Secondary | FAS | MMRM | - | - |

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 2 April 2021 1.0 Final 21 of 25

12 April 2021 | Novo Nordisk

### Analyses addressing the primary estimand

The exploratory endpoints regarding the CoEQ will be analysed using the same imputation approach as used for the primary endpoints and to address the primary estimand. The imputation model is the same as for the primary endpoints with body weight replaced by assessments of the endpoint to be analysed. The statistical model for continuous endpoints will be ANCOVA with factor and covariate as for the primary endpoint % weight change with baseline body weight replaced by the baseline assessment of the endpoint to be analysed.

Handling of missing week 104 values for the primary estimand

The imputation method RD-MI will be modified for the CoEQ item scores as follows:

- 1. Imputed values will be rounded to whole numbers.
- 2. Imputed values outside the 0-10 scale will be truncated to the nearest extreme value.

### Analysis addressing the secondary estimand

The exploratory endpoint which relate to the exploratory objective regarding the CoEQ for week 104 will be analysed to address the secondary estimand using the same MMRM for efficacy described for the primary endpoints.

### 2.3.4 Explorative statistical analysis for pharmacogenetics and biomarkers

The statistical analysis of the biomarker endpoint is described under section 10.3.2.2 of the study protocol.

### 2.3.5 Other analyses

All collected data that were not defined as endpoints will be summarised by descriptive statistics.

### 2.4 Pharmacokinetic and/or pharmacodynamic modelling

Not applicable for this trial.

### 3 Changes to the statistical analyses planned in the protocol

The main analyses were described in the protocol for the trial NN9536-4378. However, clarifications and more detailed descriptions of endpoints and analyses are provided in this SAP. The changes from the protocol of NN9536-4378 are summarised below:

### 3.1 Trial-specific changes

- The CoEQ will be analysed statistically using both the primary estimand and the hypothetical estimand for the 19 items and 4 domains from baseline to week 104.
- The supportive secondary endpoint "Body weight reduction ≥ 20% from baseline at week 0" was added both for week 52 and 104.
- The statement "The comparison will be done using the primary estimand at week 52 and week 104" was deleted as the secondary estimand will cover all affect-related objectives.

Statistical Analysis Plan Trial ID: NN9536-4378 UTN:U1111-1202-1740 EudraCT No.:2017-003726-32


Date: Version: Status: Page: 2 April 2021 1.0 Final 22 of 25

12 April 2021 | Novo Nordisk

### 3.2 Changes applied across STEP trials

- The text "rescue intervention" was replaced with "anti-obesity therapies" in the estimand definitions in order to avoid any potential confusion with diabetes rescue medication.
- It has been corrected that the secondary estimand will cover all effect-related objectives.
- It was clarified that subjects in the FAS/SAS will be evaluated "as randomised"/"as treated".
- In the text describing that "In general, the on-treatment period will therefore be from the date of first trial product administration to date of last trial product administration" the following has been added "(+14 days)" to emphasize that the lag-time after last trial product administration is included in the on-treatment period.
- The text explaining how to handle missing baseline values has been changed to make it clear that if no eligible observation at or before randomisation is available then the mean of baseline values across all subjects is used as baseline value.
- All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) coding.
- The BMI-grouping "27-<35" has been changed to "-<35", since subjects may lose weight between the screening and the randomisation visit, and therefore have a BMI below 27 kg/m<sup>2</sup> at the time of randomisation.
- It is clarified that RD-MI imputation is performed according to the timing of last available observation *during the on-treatment period* (LAO-OT). This is true for all endpoints. This is to clarify that the grouping of subjects according to timing is as in McEvoy1. Furthermore it is clarified that the LAO-OT must be prior to the landmark visit (week 104).
- In grouping of retrieved subjects by timing of LAO-OT in the RD-MI procedure, it is clarified that timing by quarters or halves is defined as too restrictive if the imputation model cannot be fit due to inadequate numbers of retrieved subjects in 1 or more groups. Furthermore it is described how a model reduction will be performed if needed.
- It is clarified that if no post-baseline LAO-OT exist, then the LAO-OT will be the baseline value and the timing of LAO-OT will be the first interval.
- In all multiple imputation procedures, in addition to the seed number, it is specified that the dataset is sorted by subject ID.
- The TP-MI procedure has been updated to be a 2-way tipping point analysis in which penalties are applied to both treatment groups (semaglutide 2.4 mg and placebo).
  - First, missing data are imputed according to the primary multiple imputation approach. Then, a penalty is added to the imputed value at week 104. The approach is to explore a range of penalties for both treatment groups, and the impact these have on the study conclusions. The 2-dimensional space of penalties covering the range from -30% to 30% will be explored for both treatment groups. This sensitivity analysis evaluates the robustness of the superiority conclusions to departures from the observed change in body weight in both treatment groups.
  - O The rationale for the change in TP-MI is the following feedback from FDA: "To confirm the robustness of superiority conclusions using a tipping point analysis, we believe that a 2-way tipping point analysis represents the real-world situation for missing data from the both treatment arms (semaglutide and placebo). We would like to see departures from the treatment difference by varying both treatment arms rather than only adding a penalty to the active treatment arm (semaglutide).

| Statistical Analysis Plan<br>Trial ID: NN9536-4378<br>UTN:U1111-1202-1740<br>EudraCT No.:2017-003726-32 | CONFIDENTIAL | Date:<br>Version:<br>Status:<br>Page: | 12 April 2021<br>1.0<br>Final<br>23 of 25 | Novo Nordisk |
|---|---|---|---|---|
|---|---|---|---|---|

Additionally, please include interpretations for the varying scenarios and how likely they would be seen in a real-world setting".

- A description has been included of the sensitivity analysis of the 5% responder endpoint (primary estimand) using MMRM.
- It has been clarified that the non-responder analysis includes subjects with missing body weight assessment at week 104 as non-responders.
- It has been clarified that the 5% responder analysis using MMRM for the secondary estimand will be predicting individual values for body weight only when body weight is missing at week 104. Furthermore, it is clarified that the logistic regression will include both randomised treatment as a factor and baseline body weight as covariate.
- It is specified that fasting serum insulin will be log-transformed and analysed using a multiplicative model.
- It is specified that lipids, FPG and fasting insulin will also be analysed in SI-units.

 Statistical Analysis Plan
 Date:
 12 April 2021
 Novo Nordisk

 Trial ID: NN9536-4378
 Version:
 1.0
 1.0

 UTN:U1111-1202-1740
 Status:
 Final

 EudraCT No.:2017-003726-32
 Page:

### 4 Change log

### SAP change log

| Version | Reason for change |
|---------|-------------------|
| 1.0 | New |

 Statistical Analysis Plan
 Date:
 12 April 2021
 Novo Nordisk

 Trial ID: NN9536-4378
 Version:
 1.0
 1.0

 UTN:U1111-1202-1740
 Status:
 Final

 EudraCT No.:2017-003726-32
 Page:

### 5 References

- 1. McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6.
- 2. Carpenter JR, Roger JH, Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat. 2013;23(6):1352-71.
- 3. Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, et al. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009;360(9):859-73
- 4. Dalton, M., Finlayson, G., Hill, A., & Blundell, J. (2015). Preliminary validation and principal components analysis of the Control of Eating Questionnaire (CoEQ) for the experience of food craving. European Journal of Clinical Nutrition, Vol. 69, p. 1313-1317.